CLINICAL TRIAL: NCT03774550
Title: A Comparison of Radiofrequency Catheter Ablation With or Without Contact-force and Cryoablation for Paroxysmal Atrial Fibrillation Ablation
Brief Title: Atrial Fibrillation Ablation: Radiofrequency or Cryoablation?
Acronym: ARCFA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-05Obs-CHRMT
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Catheter ablation; Radiofrequency; Contact-force; Cryoablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to compare 3 techniques routinely used for paroxysmal atrial fibrillation ablation: radiofrequency catheter ablation without contact-force, radiofrequency catheter ablation with contact-force and cryoablation. The hypothesis is the non-inferiority between the 3 techniques in terms of free-from atrial fibrillation survival (primary criteria). It will also compare lenght of procedure, radioscopy time and immediate complications (secondary criteria).

ELIGIBILITY:
Inclusion Criteria:

* Patients who had an atrial fibrillation for symptomatic paroxysmal atrial fibrillation, refractory to antiarrhythmic drugs, between 01/01/2014 and 30/09/2017 in CHR Metz-Thionville

Exclusion Criteria:

* Patients not willing to participate via using their medical files

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had an atrial fibrillation for symptomatic paroxysmal atrial fibrillation, refractory to antiarrhythmic drugs, between 01/01/2014 and 30/09/2017 in CHR Metz-Thionville
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation survival | Day 1
  Free from atrial fibrillation survival

SECONDARY OUTCOMES:
Immediate complications | Day 1
  The number of immediate complications encountered
Radioscopy duration | Day 1
  Radioscopy duration
Lenght of procedure | Day 1
  Overall duration of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, Moselle, France